CLINICAL TRIAL: NCT00539227
Title: A Pilot Study to Evaluate Nipple-Areolar Complex (NAC) Sparing Mastectomy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0194
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Nipple-Areolar Complex; Mastectomy; Prophylactic mastectomy; Immediate reconstruction; Reconstructive surgery; Questionnaire; Survey; NAC
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NAC Sparing Mastectomy: A skin-sparing mastectomy performed with preservation of the nipple-areolar complex (NAC). Questionnaires taking about 20-30 minutes to complete.
  Interventions: Procedure: NAC Sparing Mastectomy; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: NAC Sparing Mastectomy — A skin-sparing mastectomy performed with preservation of the nipple-areolar complex (NAC).
Behavioral: Questionnaire — Questionnaires taking about 20-30 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this study is to study nipple-areolar complex (NAC) sparing mastectomy as an alternative procedure to the standard skin-sparing mastectomy for women who have breast cancer or are at high-risk for developing breast cancer. You have been asked to take part in this study because your treating surgeon feels you are a candidate for skin-sparing mastectomy and because you want breast reconstruction after surgery. Outcomes that will be measured include how much nipple sensation can be kept after surgery; how satisfied you are with how the breast looks after surgery; complication rates; and your quality-of-life.

DETAILED DESCRIPTION:
Operative Procedure:

You will have a skin-sparing mastectomy performed with preservation of the NAC. During surgery, the tissue will be tested while you are still under general anesthesia.

The NAC may be removed completely during the surgery if malignant cells are found during the testing done during the surgery or if suspicious cells that are not clearly benign cells are found. This will be up to your doctor. The NAC may also be removed surgically if the primary tumor is found to be located less than an inch from the border of the NAC, or you are found to have breast cancer with multiple "center" sites. The nipple can also be removed by itself, with the areola spared (this is called "areolar-sparing mastectomy") if your doctor is worried about its blood supply. These decisions will be made by your pathologist and treating surgeon.

You will then undergo immediate reconstruction, with either your own tissue, prosthetic tissue, or a combination of the two. This is up to your plastic surgeon. You will have met with your plastic surgeon before surgery to discuss the best reconstructive method for you, and you will be given an informed consent to sign at that time with details about the method you decide to use.

The breast tissue under the NAC will be biopsied and tested after your surgery. After that tissue has been tested, a second surgery may be needed if cancer cells are found, the tumor is too close to the NAC, or it has more than 1 "center" site. You will have the whole NAC removed in a separate operation. The place where the NAC was removed will be repaired by a plastic surgeon, who will choose the best method to get an acceptable cosmetic result. This may involve one or more extra surgeries, and you will be given separate informed consent documents to sign for each surgery.

Follow-up and Questionnaires:

If you agree to take part in this study, 4 sensory tests will be conducted on both breasts using a variety of hand-held devices. These tests are painless and will be performed at regularly scheduled follow-up visits in clinic. They will measure nipple and areolar sensitivity, as well as nipple erectibility. The tests will involve the placement of fibers of various thicknesses and blunt metal probes on the skin of your nipple and areola. All tests will be performed once before the surgery and then at about 3 months, 6 months, and 1 year after surgery, at your follow-up clinic visits.

Your breasts will be photographed at your 6-month and 1-year follow-up visits after surgery. At these visits, you will look at those photographs to decide how satisfied you are with how the breasts look. Two (2) plastic surgeons not directly involved in your surgery will also study those photographs by themselves and fill out a similar questionnaire rating their impression of the results of your plastic surgery. These results will not be made available to you. You will also complete 2 quality-of-life questionnaires within 1 month of your surgery, and then at 3 months, 6 months, 1 year, 2 years, and 5 years after surgery (+/- 1 month). The questionnaires will ask questions about nipple sensation, cosmetic outcomes, complications, and your quality of life. The questionnaires will take about 30 minutes to complete.

Length of Study:

You will remain on study for up to 5 years.

This is an investigational study. Up to 37 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients desiring prophylactic mastectomy with immediate reconstruction
2. Patients with Stage 0, I, or II breast cancer who are candidates for and desire skin-sparing mastectomy with immediate reconstruction
3. Tumor location greater than or equal to 2.5 cm from the border of the NAC based on preoperative imaging and/or clinical exam
4. Patients must sign an informed consent and be registered before the procedure is performed

Exclusion Criteria:

1. Patients with cancer involvement of the NAC on clinical exam, defined as induration, retraction, fixation, ulceration, or pathologic nipple discharge
2. Patients with subareolar tumor locations, tumors located < 2.5 cm from the border of the NAC
3. Patients with Paget's disease of the nipple
4. Patients who have locally advanced breast cancer manifesting as inflammatory breast cancer or gross involvement of the mastectomy skin
5. Patients with history of prior surgery involving a periareolar incision
6. Patients desiring a concomitant ipsilateral reduction mammoplasty at time of mastectomy
7. Patients with macromastia as defined by the plastic surgeon
8. Patients with a body mass index (BMI) greater than 40 kg/m2
9. Patients who actively smoke
10. Patients with known collagen vascular disease
11. Patients with prior ipsilateral chest wall irradiation less than 12 months from their time of surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2007-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Nipple Sensation Evaluation (following NAC sparing mastectomy) | Within first month postoperatively, then at 3 months, 6 month, 1 year, 2 years, and 5 years postoperatively (each interval +/- 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Gildy V. Babiera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org